CLINICAL TRIAL: NCT05095246
Title: A Phase I Study of Inhaled KB407, a Replication-Incompetent, Non-Integrating Vector Expressing Human Cystic Fibrosis Transmembrane Conductance Regulator (CFTR), for the Treatment of Cystic Fibrosis
Brief Title: A Study of Inhaled KB407 for the Treatment of Cystic Fibrosis
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Pandemic, logistical, and recruitment challenges
Sponsor: Krystal Biotech, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KB407-01
Record Dates: First submitted 2021-08-27; First posted 2021-10-27 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (KB407) (Experimental): A single dose of KB407 administered on Day 0
  Interventions: Biological: KB407 (Nebulization)
- Cohort 2 (KB407) (Experimental): Two (2) doses of KB407 administered at Day 0 and Day 14
  Interventions: Biological: KB407 (Nebulization)
- Cohort 3 (KB407) (Experimental): Four (4) doses of KB407 administered at Day 0, Day 7, Day 14, and Day 21
  Interventions: Biological: KB407 (Nebulization)

INTERVENTIONS:
Biological: KB407 (Nebulization) — Nebulized solution of KB407, a replication-incompetent HSV-1 expressing full length human CFTR

SUMMARY:
The Sponsor is developing KB407, a replication-defective, non-integrating herpes simplex virus type 1 (HSV-1)-derived vector engineered to deliver functional full-length human Cystic Fibrosis Transmembrane Conductance Regulator (CFTR) to the airways of people with cystic fibrosis via nebulization. This study is designed to evaluate safety and tolerability of KB407 in people with cystic fibrosis. This study will enroll 4 participants into each of the first two cohorts and will enroll five subjects into the last cohort. Cohort 1 will receive a single dose of KB407 and be followed for 60 days. Subjects in Cohort 1 may rollover into Cohort 2 at the Day 28 Visit. A Data Safety Monitoring Board (DSMB) will meet to determine study progress from Cohort 2 into Cohort 3. In Cohort 2, subjects will be dosed bi-weekly at Day 0 and Day 14. In Cohort 3 subjects will be dosed weekly at Day 0, Day 7, Day 14 and Day 21. All subjects will be followed for a year after the last dose of KB407.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or legally appointed and authorized representative must have read, understood and signed an Institutional Review Board/Ethics Committee (IRB/EC) approved Informed Consent Form and must be able to and willing to follow study procedures and instructions.
2. Male or female subject aged 18 years old or older at the time of Informed Consent.
3. A confirmed diagnosis of cystic fibrosis (CF) that is clinically stable, in the opinion of the Investigator.
4. FEV1 ≥50% and ≤100% of the predicted normal for age, gender, and height at Visit 1 (Screening).

Exclusion Criteria:

1. Initiation of any new chronic therapy (e.g., ibuprofen, hypertonic saline, azithromycin, Pulmozyme®, Cayston®, TOBI®) or any change in chronic therapy (excluding pancreatic enzyme replacement therapy) within 28 days of Visit 2 (Day 0).
2. Hospitalization, sinopulmonary infection, CF exacerbation, or other clinically significant infection or illness within 14 days of Visit 2 (Day 0) that, in the opinion of the Investigator, may confound study results.
3. A positive culture (saliva or sputum) indicating infection with highly virulent bacteria associated with accelerated decline in pulmonary function and/or decreased survival (e.g., Burkholderia cenocepacia, Burkholderia dolosa, Mycobacterium abscessus) within 6-months of Visit 2 (Day 0).
4. Participation in another clinical study or treatment with an investigational agent within 30 days or 5 half-lives, whichever is longer, of Visit 2 (Day 0).
5. History of lung transplantation.
6. Any condition (including a history or current evidence of substance abuse or dependence) that, in the opinion of the Investigator, would impact a subject's ability to complete all study-related procedures and/or poses an additional risk to the assessment of safety of the Investigational Product (IP).
7. An active oral herpes infection within 30 Days of Visit 2 (Day 0).
8. Women who are pregnant or nursing.
9. Subject who is unwilling to comply with contraception requirements per-protocol.
10. Clinically significant abnormalities of hematology or chemistry testing at Visit 1 (Screening) that the Investigator believes may interfere with the assessment of safety and/or efficacy of the study treatment.
11. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of KB407 in subjects with Cystic Fibrosis through adverse events as assessed by NCI-CTCAE v5.0 | Baseline to End of the treatment assessed up to an average of 60 days
  Number of participants with treatment related adverse events as assessed by NCI-CTCAE v5.0

SECONDARY OUTCOMES:
To measure the difference in lung function over the course of the study, by change from baseline in forced expiratory volume (FEV1). | Baseline to End of the treatment up to an average of 60 days
  Assessment of forced expiratory volume, in one second (FEV1,) will be assessed by pulmonary function test (PFT) as compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Medical Research Institute, Newcastle, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No